CLINICAL TRIAL: NCT06810349
Title: A Multicenter Study on Predicting Tumor Origin Based on Deep Learning of Lymph Node Puncture Cytology
Brief Title: Predicting Tumor Origin Based on Deep Learning of Lymph Node Puncture Cytology
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jianyong Lei, Professor, West China Hospital
Other Study IDs: 2024 Audit No. (1041)
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Lymph Nodes With Tumor Metastasis
Keywords: Primary unknown tumor origin; Deep learning; Cytopathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Lymph node aspiration cytology imaging data
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- a training cohort and a validation cohort: Training cohort: Lymph node cytology smear imaging data and corresponding clinical data from October 1, 2008-August 31, 2024 in West China Hospital of Sichuan University.
  Validation cohort: Lymph node cytology smear imaging data and corresponding clinical data from January 1, 2020-August 31, 2024 in the First Affiliated Hospital of Zhengzhou University, Sichuan Provincial Cancer Hospital, and the Cancer Hospital of China Academy of Medical Sciences.

SUMMARY:
In this study, the investigators aimed to construct a deep learning diagnostic model that uses cytological images to predict primary unknown tumor origins in patients with tumors combined with lymph node metastases. After the model is constructed, the model will be validated by a large-scale test set to test the model performance. The investigators also propose to compare the performance of the constructed model in diagnosing cytology smears compared to human pathologists.

ELIGIBILITY:
Inclusion Criteria:

* From West China Hospital of Sichuan University (October 1, 2008-August 31, 2024) with corresponding clinical data, including age, sex, specimen puncture site, pathologic diagnosis, pathologic type, whether immunocytochemistry was added, clinical diagnosis, lesion site, co-morbidities, history of malignancy, treatment modality, occurrence of postoperative complications, total number of days of hospitalization postoperatively, and survival time;
* From the Department of Pathology of the First Affiliated Hospital of Zhengzhou University, the Sichuan Provincial Cancer Hospital, and the Cancer Hospital of the Chinese Academy of Medical Sciences (January 1, 2020-August 31, 2024) with corresponding clinical data, including age, sex, specimen puncture site, pathologic diagnosis, pathologic type, whether immunocytochemistry was added, clinical diagnosis, lesion site, co-morbidities, history of malignancy, treatment modality, occurrence of postoperative complications, total number of days of hospitalization postoperatively, and survival time.

Exclusion Criteria:

* Images lacking any supporting clinical or pathologic evidence to support a primary origin and its corresponding clinical information;
* Blank, poorly focused, and low-quality images containing severe artifacts and their corresponding clinical information.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Lymph node cytology smear imaging data and clinical data in the training cohort were obtained from West China Hospital of Sichuan University (October 1, 2008 to August 31, 2024).
  Lymph node cytology smear imaging data and clinical data in the validation cohort were obtained from the Department of Pathology of the First Affiliated Hospital of Zhengzhou University, Sichuan Cancer Hospital, and Cancer Hospital of the Chinese Academy of Medical Sciences (January 1, 2020 to August 31, 2024).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Model performance metrics | 1 year
  Model performance was evaluated by Positive Predictive Value (PPV), Negative Predictive Value (NPV), Accuracy, Sensitivity and Specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
The availability of the large amount of cytology image imaging data from the study is limited due to its oversized storage and therefore not publicly available.